CLINICAL TRIAL: NCT04334174
Title: A Phase II Single Arm Proof of Concept, Safety, Efficacy, Multicenter Study of Brentuximab Vedotin as Consolidation Therapy After Autologous Stem Cell Transplant in CD30 Expressing Peripheral T Cell Lymphomas
Brief Title: Study of Brentuximab Vedotin as Therapy After Autologous Stem Cell Transplant in Cluster of Differentiation Antigen 30 (CD30) Positive Peripheral TCell Lymphomas
Acronym: BRENTICON-T
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: accrual not met
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Principal Investigator, Marc Hoffmann, MD, University of Kansas Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2019-BRENTICON-T
Record Dates: First submitted 2020-03-20; First posted 2020-04-06 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: T Cell Lymphoma
Keywords: CD30 Positive Mature T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Brentuximab vedotin (SGN-35), intravenous infusion, 1.8 milligrams (mg) per kilogram (kg), day one of each twenty- one day cycle with a total of ten cycles planned.
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab Vedotin will be dosed at 1.8 milligram (mg) per (/) kilogram (Kg) of participants body weight will be infused intravenously every three weeks for up to ten infusions.
  Other Names: Adcetris, SGN-35

SUMMARY:
For participants with CD30 positive Mature T-cell lymphomas who have received brentuximab vedotin, cyclophosphamide, doxorubicin, and prednisone (A-CHP) as induction (4 to 6 cycles) and achieved complete response (CR) or chemo-sensitive partial response (PR) and deemed suitable for autologous stem cell transplant (ASCT) as consolidation, the investigators propose to add brentuximab vedotin after ASCT.

There is currently no standard of care treatment to prevent relapse after upfront treatment or ASCT for CD30-positive peripheral T-cell lymphoma's (PTCL)s. An agent that could improve outcomes in this population would be a major contribution to the field and is likely to be practice changing. Therefore, in addition to studying the anti-lymphoma activity of A-CHP as induction therapy, for participants who respond to induction the investigators propose to add brentuximab vedotin consolidation after ASCT in participants treated with consolidative upfront ASCT.

ELIGIBILITY:
Inclusion Criteria:

* A-CHP for 6 cycles. First cycle may be cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP)- based if already planned and then 5 cycles of A-CHP.
* Performance status of 0-2.
* Participants with CD30 positive mature T- cell lymphomas who have received A-CHP as induction and achieved complete response (CR) or chemo- sensitive partial response (PR) and deemed suitable for ASCT as consolidation.
* Eligible disease types:

  * Anaplastic lymphoma kinase (ALK)- negative systemic Anaplastic large-cell lymphoma (sALCL)
  * Peripheral T-cell lymphoma- not otherwise specified (PTCL-NOS)
  * Angioimmunoblastic T-cell lymphoma (AITL)
  * Adult T-cell leukemia/lymphoma (ATLL; acute and lymphoma types only, must be positive for human T cell leukemia virus 1)
  * Enteropathy-associated T-cell lymphoma (EATL)
  * Hepatosplenic T-cell lymphoma (HSTCL)
* Fluorodeoxyglucose (FDG)-avid disease by positron emission tomography (PET) and measurable disease by Computed tomography (CT), as assessed by the site radiologist.
* Adequate organ function.

Exclusion Criteria:

* Enrolled in any other treatment clinical trial.
* Is breastfeeding.
* Active severe or medically significant or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of study treatment.
* Has human immunodeficiency virus (HIV) infection, hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection.
* Left ventricular ejection fraction (LVEF) less than 45% or symptomatic cardiac disease, or myocardial infarction within the past 6 months.
* Previous treatment with complete cumulative doses of doxorubicin or other anthracyclines.
* Baseline, moderate, peripheral neuropathy or patients with the demyelinating form of Charcot-Marie-Tooth syndrome.
* Post auto or allo stem cell transplant (SCT).
* Cerebral/meningeal disease related to the underlying malignancy.
* History of progressive multifocal leukoencephalopathy (PML).
* Current diagnosis of any of the following:

  * Primary cutaneous CD30-positive T-cell lymphoproliferative disorders and lymphomas. Cutaneous ALCL with tumor spread outside of the skin and to lymph nodes away from the primary site are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who experience safety related issues caused by study treatment: CTCAEv5 | Up to three years
  Using the Common Terminology Criteria for Adverse Events version 5 (CTCAEv5) to evaluate participants reaction to treatment.

SECONDARY OUTCOMES:
Progression Free Survival | From date of randomization until the date of first documented progression or to death due to any cause, whichever comes first, up to 3 years.
  Comparing statistical survival rates with survival rates of study participants.
The number of adverse events or laboratory abnormalities | 30 days
  Monitoring the number of adverse events or laboratory abnormalities using the CTCAEv5 as reference.

CONTACTS AND LOCATIONS:
Overall Officials: Sid Ganguly, MD, Principal Investigator — The University of Kansas
Locations (1):
- The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas, United States